CLINICAL TRIAL: NCT00575380
Title: A Multi-Center, Open-Label, Randomized Study of the Pharmacokinetics of Azithromycin Versus Moxifloxacin in Conjunctiva and Aqueous Humor Following Single or Multiple Ocular Administration of AzaSite Ophthalmic Solution, 1% or Vigamox in Subjects Undergoing Routine Cataract Surgery
Brief Title: Study of AzaSite Versus Vigamox Concentrations in the Conjunctiva and Aqueous Humor in Subjects Undergoing Routine Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Mike Schiewe, Inspire Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 041-103; P08655
Record Dates: First submitted 2007-12-12; First posted 2007-12-18 (Estimated); Results first posted 2009-09-16 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Bacterial Infections; Eye Infections; Cataract Extraction
MeSH Terms: conditions — Bacterial Infections; Eye Infections | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AzaSite Eye Drops (Active Comparator): One drop two times a day for two days and once a day for the next five days
  Interventions: Drug: AzaSite Eye Drops
- Vigamox Eye Drops (Active Comparator): One drop three times a day for seven days
  Interventions: Drug: Vigamox Eye Drops

INTERVENTIONS:
Drug: AzaSite Eye Drops — One drop two times a day for two days and once a day for the next five days.
  Other Names: AzaSite (azithromycin ophthalmic solution)
  Arms: AzaSite Eye Drops
Drug: Vigamox Eye Drops — One drop three times a day for seven days
  Other Names: Vigamox(moxifloxacin hydrochloride ophthalmic solution)
  Arms: Vigamox Eye Drops

SUMMARY:
The purpose of this study is to evaluate the drug concentrations in the conjunctiva and aqueous humor of AzaSite™ compared to Vigamox® in subjects undergoing routine cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Are scheduled to undergo routine cataract surgery by the investigator's preferred technique.
* Have normal appearing, freely mobile, conjunctiva in the inferior temporal portion cul-de-sac site of the operative eye.

Exclusion Criteria:

* Have concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye.
* Have a history of ocular pemphigoid.
* Have ever had penetrating ocular surface surgery.
* Have had intraocular surgery within the past 3 months.
* Have ever had prior surgery or full penetrating trauma to the conjunctiva at the proposed surgical site.
* Have a planned cataract surgery in the contraleteral eye within 2 weeks of the study related surgical procedure and sample collection.
* Have a combined procedure planned (trabeculectomy surgery planned in the same eye as cataract extraction surgery).
* Have at the proposed conjunctiva biopsy site, signs of conjunctival shortening of the fornix, scarring or adherence to the underlying episclera.
* Have according to the investigator's judgment, risk of intra- or post-operative complications related to their cataract surgery as a consequence of participation in the study.
* Have a known hypersensitivity to azithromycin, or any macrolide antibiotic or to any of the ingredients in AzaSite.
* Have had a known hypersensitivity to Vigamox or any fluoroquinolone antibiotics or to any of the ingredients in Vigamox.
* Are unable or unwilling to withhold for a minimum of 3 weeks prior to initiation of study drug, the ocular or systemic use of either azithromycin or moxifloxacin, when it is the same medication as the subject's assigned study drug. This relates as well, to the use of either of these medications as a pre-surgical prophylaxis.
* Are unable or unwilling to withhold for a minimum of 3 weeks prior to initiation of study drug, the use of erythromycin ointment or ofloxacin.
* Have any ocular pathology with the exception of cataracts that in the judgment of the investigator could confound study assessments or limit compliance.
* Have a serious systemic disease or uncontrolled medical condition or psychiatric condition that in the judgement of the investigator could confound study assessments or limit compliance.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- United States (13):
  - Cornea Consultants of Arizone, Phoenix, Arizona
  - Eye Care Arkansas, Little Rock, Arkansas
  - North Valley Eye Medical Group, Mission Hills, California
  - Center for Excellence in Eye Care, Miami, Florida
  - Eye Center of North Florida, Panama City, Florida
  - Coastal Research Associates, LLC, Atlanta, Georgia
  - Kentuckiana Institute for Eye Research, Louisville, Kentucky
  - Ophthalmology Associates, St Louis, Missouri
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Eye Care Specialists, Kingston, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Glaucoma Consultants and Center for Eye Research, Mt. Pleasant, South Carolina
  - Corona Research Consultants, El Paso, Texas

REFERENCES:
- [Derived] Stewart WC, Crean CS, Zink RC, Brubaker K, Haque RM, Hwang DG. Pharmacokinetics of azithromycin and moxifloxacin in human conjunctiva and aqueous humor during and after the approved dosing regimens. Am J Ophthalmol. 2010 Nov;150(5):744-751.e2. doi: 10.1016/j.ajo.2010.05.039. Epub 2010 Sep 1. PMID 20813346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azasite | Vigamox
Started | 58 | 58
Completed | 57 | 55
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Various | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azasite | Vigamox | Total
Number analyzed (Participants) | 58 | 58 | 116
Age Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.57) | 66.3 (10.02) | 68.6 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 62
  Male | 24 | 30 | 54

OUTCOME MEASURES:

1. Primary Outcome: Conjunctiva Concentration Prior to Cataract Surgery at One of Ten Time Points Ranging From 1 to 14 Days (Per Protocol Pharmacokinetic Population)
Description: Nominal time is scheduled time relative to administration of the first eye drop
Time Frame: Az(hr): 1,12,48,49,72,144,145,168,216,312; Vig(hr): 1,8,48,49,56,144,145,168,216,312
Measure: Mean (Standard Deviation); unit: ug/g
Arm/Group | Azasite | Vigamox
Number analyzed (Participants) | 57 | 55
ug/g
  Timepoint 1 - 1 hr (AzaSite and Vigamox) | 40.4 (19.7752) | 5.747 (3.4775)
  Timepoint 2 - 12 hrs (AzaSite)/8 hrs (Vigamox) | 33.55 (11.81) | 1.051 (.8099)
  Timepoint 3 - 48 hrs (AzaSite and Vigamox) | 559.733 (1011.658) | 1.129 (1.1673)
  Timepoint 4 - 49 hrs (AzaSite and Vigamox) | 98.6 (4.535) | 15.754 (15.4107)
  Timepoint 5 -72 hrs (AzaSite)/56 hrs (Vigamox) | 287.75 (433.4355) | .862 (.6801)
  Timepoint 6 - 144 hrs (AzaSite and Vigamox) | 175.017 (88.9250) | .305 (.0917)
  Timepoint 7 - 145 hrs (AzaSite and Vigamox) | 269.46 (316.2821) | 5.432 (4.0756)
  Timepoint 8 - 168 hrs (AzaSite and Vigamox) | 261.125 (169.1224) | .322 (.1792)
  Timepoint 9 - 216 hrs (AzaSite and Vigamox) | 273.9 (160.4984) | .165 (.1974)
  Timepoint 10 - 312 (AzaSite and Vigamox) | 63.867 (51.1578) | .011 (.0098)

2. Secondary Outcome: Aqueous Humor Concentration Prior to Cataract Surgery at One of Ten Time Points Ranging From 1 to 14 Days (Per Protocol Pharmacokinetic Population)
Time Frame: Az(hr): 1,12,48,49,72,144,145,168,216,312; Vig(hr): 1,8,48,49,56,144,145,168,216,312
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Azasite | Vigamox
Number analyzed (Participants) | 57 | 55
ug/mL
  Timepoint 1- 1 hr (AzaSite and Vigamox) | .022 (.0297) | .582 (.506)
  Timepoint 2- 12 hrs (AzaSite)/ 8 hrs (Vigamox) | .088 (.0084) | .113 (.0729)
  Timepoint 3 - 48 hrs (AzaSite and Vigamox) | .047 (.0515) | .079 (.0543)
  Timepoint 4 - 49 hrs (AzaSite and Vigamox) | .023 (.0183) | .765 (.5657)
  Timepoint 5 - 72 hrs (AzaSite)/ 56 hr (Vigamox) | .02 (.0099) | .084 (.0261)
  Timepoint 6 - 144 hrs (AzaSite and Vigamox) | .026 (.0175) | .225 (.1456)
  Timepoint 7 - 145 hrs (AzaSite and Vigamox) | .052 (.0694) | .669 (.402)
  Timepoint 8 - 168 hrs (AzaSite and Vigamox) | .035 (.0276) | .059 (.0265)
  Timepoint 9 - 216 hrs (AzaSite and Vigamox) | .028 (.0353) | .071 (.0845)
  Timepoint 10 - 312 hrs (AzaSite and Vigamox) | .011 (.0102) | .017 (.0189)

ADVERSE EVENTS:
Arm/Group | Azasite | Vigamox
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 3/58 | 2/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azasite (N=58) | Vigamox (N=58)
Intraocular pressure increased (Investigations) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish or discuss trial results until written communication is received from Inspire